CLINICAL TRIAL: NCT06789783
Title: Cornelia De Lange Syndrome: Assessing Positive Effects of Lithium Treatment
Acronym: CLoSER
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Aglaia Vignoli, Professor, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210-18042023; patients association (Other: ASST Niguarda)
Record Dates: First submitted 2024-12-19; First posted 2025-01-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Cornelia De Lange Syndrome
Keywords: Lithium treatment
MeSH Terms: conditions — De Lange Syndrome | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CdLS patients with NIPBL mutation (Experimental): Patients will be given 10mg/Kg twice a day, 150mg or 300mg Lithium Carbonate
  Interventions: Drug: Lithium Carbonate Capsule

INTERVENTIONS:
Drug: Lithium Carbonate Capsule — 10mg/Kg twice a day, 150mg or 300mg Lithium Carbonate

SUMMARY:
The study "Cornelia de Lange Syndrome: assessing positive effects of Lithium treatment - CLoSER" aims to evaluate the effectiveness on behavioral modifications of lithium carbonate therapy in patients with Cornelia de Lange syndrome (CdLS).

CdLS is a rare genetic disease caused by autosomal mutations dominant or X-linked. The prevalence of CdLS is estimated to be between 1:10,000-30,000 newborns, but it is probably underestimated because the most cases mild ones may go undiagnosed. This syndrome is characterized by slow growth before and after birth with intellectual disability and short stature, from major malformations such as facial anomalies, neurological disorders, gastrointestinal and musculoskeletal malformations. To date, for these patients only targeted medical and surgical therapeutic interventions are recommended for improving the quality of life. No drug therapy is validated for the cognitive/behavioral disorders. It has been shown that lihium-dependent activation of the WNT pathway is able to recover the Abnormal phenotype in many CdLS models. Lithium is already widely used in psychiatry and has a long history of clinical efficacy.

Recently some studies are evaluating the effect of lithium in patients with characteristics common to CdLS showing promising results . This trial intends to transfer the preliminary data obtained from in vitro and in vivo studies on patients with CdLS.

Given the currently untreatable nature of the syndrome, this treatment could represent a possible therapeutic strategy aimed at improving the behavioral and intellectual disabilities typical of CdLS.

DETAILED DESCRIPTION:
Research Objectives This study aims to evaluate the effectiveness of lithium carbonate therapy on behavioral changes in patients with Cornelia de Lange syndrome (CdLS). This is a multicenter and non-commercial pilot clinical study.

The specific objectives are the following:

PRIMARY OUTCOME - Improvement in the following parameters:

• Behavior assessed by Aberrant Behavior Checklist (ABC scale1), which measures psychiatric symptoms and behavioral disorders also in patients with intellectual disability;

SECONDARY OUTCOMES - Improvement in the following parameters:

* SCQ questionnaire (SCQ; Rutter, Bailey&Lord, 20032) to assess communication skills and social functioning;
* Childhood Autism Rating Scale (CARS 2 -T3) to assess autistic behaviors;
* Cognitive Performance through the Leiter scale (Leiter-R, Roid & Miller, 19974), a non-verbal scale that can be used for subjects between 2 and 20 years old.
* Vineland Adaptive Behavior Scales 2 to evaluate adaptive functioning in the different areas (motor, communication, autonomy, socialization). For severe patients, where a direct evaluation with the Leiter may be insignificant or impossible to conduct, it would provide an adaptation quotient (AQ).
* Sleep quality through the Sleep Disturbances Scale for children (SDSC5), to be administered to parents; there are two versions, one for subjects between 6 and 16 years old, the other for children 3-6 years old;
* Impression of Change Clinical Global Impression of Change (CGI-C) completed by the clinician at each visit;
* Improvement in quality of life through Pediatric Quality of Life Inventory (PedsQL6)
* Specific biomarkers will be used to measure lipid peroxidation in cell extracts, tissues and biological fluids.

Background Cornelia de Lange syndrome (CdLS) is a rare genetic disorder caused by autosomal dominant or X-linked mutations. The prevalence of CdLS is estimated to be 1:10,000-30,000 newborns, but it is probably underestimated because milder cases may not be diagnosed. This syndrome is characterized by slow growth before and after birth with intellectual disability and short stature, major malformations such as facial anomalies, neurological disorders, and gastrointestinal and musculoskeletal malformations. Peculiar facial anomalies include arched and fused eyebrows on the midline, long eyelashes, anteverted nostrils, a mouth with downturned corners, and a very thin upper lip. To date, only medical and surgical therapeutic interventions to improve quality of life are recommended for these patients. No pharmacological therapy is validated for cognitive/behavioral disorders. Approximately 80% of patients with CdLS have mutations in one of the following 5 genes: NIPBL (60%), SMC1A, SMC3, RAD21 and HDAC8. These genes encode structural or accessory proteins of the cohesin complex. The cohesin complex is a multimeric system, highly conserved throughout cellular evolution from the most primitive life forms to human cells. Cohesins are essential elements for the structural maintenance of chromosomes (SMC) and interact with chromatin modulating its organization. Cohesins mediate the segregation of sister chromatids and play a fundamental role in the control of gene expression. A signaling pathway involved in all steps of central nervous system (CNS) development is the WNT pathway. Some of our previous studies have shown that an alteration of CNS development is related to a defect in the canonical WNT pathway. Current evidence suggests that CdLS malformations result from downregulation of molecular pathways during embryonic development and, in this context, our and previous studies have demonstrated that the canonical WNT pathway is perturbed. WNT has also recently been shown to play a key role in the functions of the cohesin complex in CdLS models and patient-derived fibroblasts. Our studies have highlighted how inhibition or loss of function of cohesins in in vivo models of CdLS affects CNS development. The WNT signaling pathway is involved in numerous events in the development and maintenance of adult tissue homeostasis by regulating cell proliferation, differentiation (including stem cell proliferation), migration, genetic stability and apoptosis, as well as in maintaining adult stem cells in a pluripotent state. LiCl-dependent activation of the WNT pathway is able to rescue the affected phenotype in CdLS models. Lithium is already widely used in psychiatry and has a long history of clinical efficacy as the first drug used in the treatment of mental illness. This drug is approved for the treatment of bipolar disorder because of its ability to stabilize mania and depression. Its use must be properly monitored so that ideal blood concentrations are maintained (0.4-1.2 mEq/L) and to monitor possible side effects. Recently, some studies have evaluated the effect of lithium in patients with features common to CdLS. A clinical trial proposed lithium therapy for the treatment of Fragile X Syndrome showing promising results. These patients exhibit traits similar to those of CdLS patients, particularly intellectual disabilities and autism spectrum disorders. Another study demonstrated the efficacy of lithium treatment as a mood stabilizer in two patients with SHANK3 gene mutations who were diagnosed with autism spectrum disorder in childhood. The project the investigators present aims to transfer the preliminary data obtained from in vitro and in vivo studies to patients with CdLS.

Due to the currently untreatable nature of the syndrome, this treatment could represent a potential therapeutic strategy aimed at improving the behavioral and intellectual disabilities commonly associated with CdLS.

Study Design the investigators designed a 52-week prospective treatment study to evaluate the efficacy of lithium carbonate in CdLS

Study Centers and Number of Subjects The investigators plan to enroll at least 34 subjects with CdLS, affiliated with the Child and Adolescent Neuropsychiatry Unit of the ASST Grande Ospedale Metropolitano Niguarda in Milan, the Pediatrics Unit of the ASST Lariana and the Child and Adolescent Neuropsychiatry Operating Unit (UONPIA) Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico in Milan. Laboratory analyses for monitoring pharmacological treatment will be performed at the laboratories of the ASSTs involved in the study according to clinical practice. Monitoring of lipid peroxidation levels for research purposes will be performed in the Applied Biology laboratories at the Department of Health Sciences, University of Milan, with funding from Prof. Valentina Massa.

Patient recruitment Subjects who meet the defined inclusion and exclusion criteria will be recruited, after signing the informed consent, at the Child and Adolescent Neuropsychiatry Unit of the ASST Grande Ospedale Metropolitano Niguarda in Milan, the Pediatrics Unit of the ASST Lariana and the Child and Adolescent Neuropsychiatry Unit (UONPIA) Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico in Milan.

Participants will receive an information document about the study and a consent form for the collection of biological material. They will also be given a telephone number and an email address to contact if they would like more information or wish to withdraw from the study for any reason.

Patients will attend the outpatient clinics of the Department of Childhood and Adolescent Neuropsychiatry (UONPIA) at the IRCSS Ca' Granda Foundation Ospedale Maggiore Policlinico in Milan for the initial NPI evaluation (T0). During the intervention period, monitoring visits will take place at the Childhood and Adolescent Neuropsychiatry unit of ASST Grande Ospedale Metropolitano Niguarda in Milan and the Pediatrics Unit of ASST Lariana at the following time points: T1, T2, T3, T4, T5, and T6.

At the end of the intervention period, participants will return to the UONPIA at the IRCSS Ca' Granda Foundation Ospedale Maggiore Policlinico of Milan (T7) to ensure continuity of care by a dedicated team of experts.

Methods The study drug, administered at a dosage of 10 mg/kg twice daily (150 mg or 300 mg lithium carbonate tablets), will be given to patients with an interval of 12 hours between doses. This proposed dosing regimen is based on previous experiences with lithium carbonate in pediatric patients. For patients who are unable to swallow capsules, the investigational medicinal product (IMP) can be provided as a solution.

The caregiver will record the date, time, and number of capsules administered on the Case Report Form (CRF). Symptoms of treatment intolerance include nausea, vomiting, diarrhea, hand tremors, fatigue, and muscle weakness. If any intolerance occurs during the study, the investigator may reduce the patient's dose, implement a single dose interruption, or switch to alternate day dosing. Patients who cannot tolerate the treatment even after a dose interruption must be withdrawn from the study.

The tapering process for treatment will involve a gradual reduction of the dosage, halving the dose every three days until complete cessation. The following medications are prohibited before and during the study:

* Concomitant antidepressants (such as venlafaxine and tricyclic antidepressants)
* Antipsychotics (including clozapine, haloperidol, phenothiazines, and risperidone)
* Antiepileptics (like carbamazepine, phenytoin, and phenobarbital)
* ACE inhibitors
* Amiodarone
* Calcium channel blockers
* Diuretics (such as thiazides and acetazolamide)
* Metronidazole
* Aminophylline
* Mannitol

Responsibilities In accordance with ICH and FDA requirements, the Investigator must always be able to account for all study drugs supplied. At the end of the study, it must be possible to reconcile the delivery records with the usage and returns records. Any discrepancies must be accounted for. Under no circumstances may the Investigator use study drugs other than those indicated in the protocol. Data collection and analysis The study will include the following phases: - Screening / Baseline (T0): subjects will be considered for the study if they meet the inclusion criteria. This phase includes: anamnesis, including drug history in treated patients and assessment of concomitant medications, and clinical assessment. Each subject will undergo cognitive assessment (Leiter-R scale and Vineland Adaptive Behavior Scales 2), behavioral scales (ABC and CARS-T) communication and social functioning scales (SCQ), sleep quality scales (SDSC) and quality of life (PedsQL) in collaboration with Dr. Ajmone of the U.O. of Childhood and Adolescent Neuropsychiatry (UONPIA) Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico di Milano. Laboratory tests (hematology, biochemistry, urinalysis, serum pregnancy test for post-pubertal females and thyroid function tests) and 12-lead ECG will be performed. In the UNIMI Applied Biology laboratory, plasma levels of TBARS, known to be associated with lithium treatment, will be assessed. Written informed consent will be collected from parents/legal representatives of eligible CdLS patients willing to participate in the study. - Start Drug Treatment (SDT, 1 week after T0): Patients included in the study start taking the drug after clinical evaluation of the tests performed at T0. Blood sampling will be performed to prepare patient-derived lymphoblastoid lines by immortalizing lymphocytes with Epstein-Barr virus (EBV) at the "Istituto Giannina Gaslini" in Genoa and the mutation of the immortalized cell lines will be confirmed using molecular genetic techniques such as PCR and Sanger sequencing at the Medical Genetics laboratory of the University of Milan. The preparation of the lines guarantees genetically characterized material on which to perform molecular and cytotoxicity assays.

* T1 (2 weeks ± 3 days after SDT): clinical evaluation, laboratory tests including serum lithium levels, thyroid and renal function and ECG. Any adverse events will be recorded and concomitant medications will be evaluated.
* T2 (2 weeks ± 3 days after T1): clinical evaluation, blood tests including serum lithium levels, thyroid and renal function and ECG, as well as safety issues.
* T3 (1 month ± 1 week after T2): Clinical evaluation, laboratory tests (hematology, biochemistry, urinalysis, serum pregnancy test for post-pubertal females, and thyroid function test), and ECG. Plasma TBARS levels will be assessed.
* T4 (1 month ± 1 week after T3): Clinical evaluation, blood tests including serum lithium level, thyroid and renal function, and ECG, as well as safety concerns.
* T5 (3 months ± 1 week after T4): Laboratory tests (hematology, biochemistry, serum lithium level, urinalysis, serum pregnancy test for post-pubertal females, and thyroid function test), and 12-lead ECG will be performed. Plasma TBARS levels will be assessed.
* T6 (3 months ± 1 week after T5) ) - end of the first study period: Laboratory tests (hematology, biochemistry, serum lithium level, urinalysis, serum pregnancy test for post-pubertal females and thyroid function tests) and 12-lead ECG will be performed. Plasma TBARS levels will be assessed.
* Follow-up T7 (3 months ± 1 week after T6): All patients will return for final assessments. A final safety level (laboratory tests, ECG, vital signs) and efficacy assessment will be performed. Baseline scales and tests will be repeated.

Patients who benefit from lithium therapy will be guaranteed continuation of treatment and related drug tolerability/safety checks. Other analyses are part of clinical practice for managing CdLS patients.

Sample size The study plan to enroll 34 patients. The sample size was calculated using the Wilcoxon test considering as a null hypothesis that there are no differences in the primary outcome parameter (ABC scale) following treatment and as an alternative hypothesis that following treatment the ABC-c value decreases by 16 points (as per clinical trial on the efficacy of lithium in patients with fragile X18) and taking into account a 10% drop out.

ELIGIBILITY:
Inclusion Criteria:

* Age > 4 years
* Body weight within the normal range in the reference range for CdLS, based on age and height
* Diagnosis of CdLS based on consensus clinical criteria and a confirmed mutation in the NIPBL gene
* Stable drug regimen for 4 weeks prior to starting the study
* Written consent signed by parent/legal guardian/representative prior to the screening visit
* Ability to take the study drug provided in capsules or drops (for younger patients and those with swallowing difficulties) or combined with food/drinks
* Caregiver must be able to understand the instructions and participate knowingly in the study

Exclusion Criteria:

* The patient is participating in another clinical trial
* QT interval prolongation, thyroid dysfunction, renal insufficiency, hepatic insufficiency, leukopenia, or other currently clinically significant medical disorders (as determined by the investigator), other than those directly related to CdLS
* QTcF interval on ECG greater than 450 msec
* Severe diabetes mellitus or inherited metabolic disorder

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Behaviour | Change at 12 months from baseline of supplementation
  Behaviour assessed through the Aberrant Behaviour checklist (ABC1 scale) which mesaure psychiatric symptomatology and behavioral disorders also in patients with intellectual disabilities. minimum total score: 0; maximum total score:174. Higher scores mean worse outcome

SECONDARY OUTCOMES:
Communication | Change at 12 months from baseline of supplementation
  Social Communication Questionnaire questionnaire (SCQ; Rutter, Bailey&Lord, 20032) to assess communication skills and social functioning; minimum score: 0; maximum score:40. Higher score means worse outcome.
Behaviour | Change at 12 months from baseline of supplementation
  Childhood Autism Rating Scale (CARS 2 -T3) to assess autistic behaviors. minimum score: 15; maximum score:60. Higher score means worse outcome. Furthermore, for very serious patients, for whom a direct assessment with the Leiter could be insignificant or impossible, it would allow for the adaptation quotient (QD).
Sleep disturbances | Change at 12 months from baseline of supplementation
  Sleep quality through the Sleep disturbances scale for children (SDSC5), to be administered to parents; there are two versions, one for subjects between 6-16 years, the other for children 3-6 years. minimum total score: 26; maximum total score:130. Higher scores mean worse outcome.
Clinical features | Change at 12 months from baseline of supplementation
  Impression of change Clinical Global Impression of Change (CGI-C) filled out by the clinician at each visit. minimum total score:0; maximum total score:30. Higher scores mean worse outcome.
Cognitive Performance | Change at 12 months from baseline of supplementation
  Cognitive Performance through the Leiter scale (Leiter-R, Roid & Miller, 19974), a non-verbal scale that can be used for subjects between 2 and 20 years old. We use only cognitive battery and administer only the 4 mandatory subtests:
  Total raw score: minimum 0, maximum 152
Adaptive functioning in the different areas | Change at 12 months from baseline of supplementation
  Vineland Adaptive Behavior Scale 2 in order to also assess adaptive functioning in the different areas (motor, communication, autonomy, socialization). minimum total score: 0; maximum total score:766. Higher scores mean better outcome
Quality of life | Change at 12 months from baseline of supplementation
  Improvement in quality of life through Pediatric Quality of Life Inventory (PedsQL6). minimum total score: 0; maximum total score:92. Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aglaia Vignoli, Professor, MD, Principal Investigator — University of Milan
Locations (1):
- University of Milan, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grazioli P, Parodi C, Mariani M, Bottai D, Di Fede E, Zulueta A, Avagliano L, Cereda A, Tenconi R, Wierzba J, Adami R, Iascone M, Ajmone PF, Vaccari T, Gervasini C, Selicorni A, Massa V. Lithium as a possible therapeutic strategy for Cornelia de Lange syndrome. Cell Death Discov. 2021 Feb 17;7(1):34. doi: 10.1038/s41420-021-00414-2. PMID 33597506